CLINICAL TRIAL: NCT04328519
Title: The Charlson Comorbidity Index: Predicting Severity in Emergency Departments
Acronym: Charlson
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Assistant Prefessor, Ataturk University
Other Study IDs: Ataturkuniversity
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Emergency Medicine
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient(hospitalized): patients who are admitted to the emergency department and hospitalized.
  Interventions: Other: observation
- control(not hospitalized): patients who are admitted to the emergency department and not hospitalized.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Objective: The Charlson Comorbidity Index (CCI) is a comorbidity scale used widely throughout the world. It uses patients' preoperative and intraoperative morbidity factors to evaluate morbidity and mortality risk. Though the CCI has widespread use, it has not been evaluated in patients attending at ES, and its relationship with patient readmission has not been shown previously. In this study, we aimed to show whether there is a correlation between the CCI value and the number of repeated admissions to emergency services and that the CCI value can be used as a predicted factor for the serious patients.

Matherials and Methods: This was a prospective observational cross-sectional study. Age, gender, vital signs of the patients who agreed to participate in the study was recorded. Numbers of emergency service applications in the last 6 months and CCI score have been recorded.

DETAILED DESCRIPTION:
This study showed that CCI score can be used for identify serious patient in emergency service.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients were told about the study, and those who agreed to participate were included

Exclusion Criteria:

* Patients who did not wish to participate in the study
* Patients who were unable to work or who had problems with consciousness
* Patients with non-hospital cardiopulmonary arrest
* Patients who had previously participated in the study (readmitted patients)
* Patients who had accessed ES for the same or a similar complaint within the last seven days
* < 18 years' old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted to the emergency room
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-07 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
determine the severity of patients. to identify patients who need hospitalization. determine the severity of patients. | 2018
  to identify patients who need hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Abdullah Osman Kocak, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No